CLINICAL TRIAL: NCT01127555
Title: Phase II Study of Salvage mFOLFOX(5-fluorouracil, Leucovorin, Oxaliplatin) in Patients With Unresectable Biliary Tract Cancer (BTC) Who Had Failed Gemcitabine
Brief Title: Salvage mFOLFOX in BTC After Failure of Gemcitabine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chung-Ang University (Other)
Collaborators: Gyeongsang National University Hospital (Other); Dong-A University Hospital (Other); Samsung Medical Center (Other)
Responsible Party: Principal Investigator, In Gyu Hwang, Chung-Ang University Hospital, Chung-Ang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAUHHO 2010-2
Record Dates: First submitted 2010-05-05; First posted 2010-05-21 (Estimated); Last update posted 2013-10-08 (Estimated); Status verified 2013-10

CONDITIONS: Unresectable Biliary Tract Cancer
Keywords: Biliary Tract Cancer; Salvage therapy; FOLFOX
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — Fluorouracil; Leucovorin; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: 5-fluorouracil, leucovorin, oxaliplatin — D1 Oxaliplatin 85mg/m2 D1, 2 LV 30mg/m2 IV push D1, 2 5-FU 1500mg/m2 CIV over 24hrs Every 2 weeks
  Other Names: mFOLFOX

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of mFOLFOX (5-fluorouracil, leucovorin, oxaliplatin)as salvage therapy in patients with unresectable biliary tract cancer who had failed gemcitabine.

ELIGIBILITY:
Inclusion Criteria:

1. Age : older than 18
2. Histologically confirmed adenocarcinoma of the biliary tract
3. Metastatic or unresectable biliary cancer
4. Prior exposure to gemcitabine chemotherapy for biliary cancer
5. Eastern Cooperative Oncology Group (ECOG) performance status 0 -2
6. A patient with at least one measurable primary lesion of which the diameter is confirmed to be 10mm in spiral Computed Tomography (CT) or multidetector CT
7. Adequate bone marrow, liver, renal function

Exclusion Criteria:

1. Pregnancy and breast-feeding.
2. Other serious illness or medical condition, notably heart or lung failure, active uncontrolled infection (infection requiring antibiotics).
3. Past or concurrent history of other neoplasm, except curatively treated basal cell skin cancer or adequately treated in-situ carcinoma of the cervix.
4. Symptomatic or uncontrolled brain metastasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-04; Primary Completion 2012-06 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Response rate | 1 year
  Clinically assessed every cycle (2weeks) and radiologically assessed every 3 cycles (6 weeks) with CT scan

SECONDARY OUTCOMES:
To evaluate the safety | 1 year
  Clinically assessed every cycle (2weeks)
To estimate the time to progression | 1 year
To estimate overall survival | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: In Gyu Hwang, M.D., Study Director — Chung-Ang University Yongsan Hospital
Locations (1):
- Chung-Ang University Yongsan Hospital, Yongsan, Seoul, South Korea